CLINICAL TRIAL: NCT02411565
Title: A Pilot Randomized, Placebo-Controlled, Trial of Fermented Wheat Germ Extract in Women With Ovarian Cancer
Brief Title: Fermented Wheat Germ Extract in Women With Ovarian Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Drug manufacturing issues
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCC-17883
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-04

CONDITIONS: Ovarian Cancer
Keywords: epithelial; ovarian; fallopian tube; primary peritoneal carcinoma; peritoneal; ovary
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Avemar; Quality of Life; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fermented Wheat Germ Extract (FWGE) (Active Comparator): FWGE administration 2 - 4 weeks prior to planned surgery, + Quality of Life (QoL) Surveys: FACT-O.
  Interventions: Drug: Fermented Wheat Germ Extract (FWGE); Other: Standard of Care: Planned Surgery; Other: Quality of Life (QoL) Surveys: FACT-O
- Placebo Administration (Placebo Comparator): Placebo administration 2 - 4 weeks prior to planned surgery, + Quality of Life (QoL) Surveys: FACT-O.
  Interventions: Drug: Placebo; Other: Standard of Care: Planned Surgery; Other: Quality of Life (QoL) Surveys: FACT-O

INTERVENTIONS:
Drug: Fermented Wheat Germ Extract (FWGE) — 5.53 grams of FWGE combined with natural orange flavor and stevia Reb-A sweetener to create an instant drink mix, dissolved in 150 mL of water, orally once-daily, for 2 to 4 weeks.
  Other Names: Avemar®
  Arms: Fermented Wheat Germ Extract (FWGE)
Drug: Placebo — Dried and pulverized, white and black rice, 5.53 grams, combined with natural orange flavor and stevia Reb-A sweetener, to create an instant drink mix, dissolved in 150 mL of water, orally once-daily, for 2 to 4 weeks.
  Arms: Placebo Administration
Other: Standard of Care: Planned Surgery — Participants will undergo their planned surgery during the 2nd to 4th week after entry into the study. However, if there are delays, patients can continue to take drug/placebo for a time period no greater than 2 months. If surgery has not occurred after this 2-month period, the patient will be removed from the study. Participants will take the study drug up until the day prior to surgery. The minimum amount of time on study drug is 2 weeks. A separate consent form will be obtained for the surgical procedure.
Other: Quality of Life (QoL) Surveys: FACT-O — Quality of life questionnaire (FACT-O) at the time of enrollment, then weekly and the day of surgery.
  Other Names: questionnaire

SUMMARY:
The main purpose of this Pilot Study is to test the safety, tolerability and quality of life in women who take Fermented Wheat Germ Extract (FWGE), to determine if an active form of FWGE can be detected in the blood, and determine whether short-term therapy with FWGE has any effect on the tumor marker, cancer antigen 125 (CA-125).

ELIGIBILITY:
Inclusion Criteria:

* Women with suspected epithelial ovarian, fallopian tube or primary peritoneal carcinoma scheduled to undergo surgical exploration with no prior treatment for the cancer. Signs of ovarian cancer include, but are not limited to: an elevated cancer antigen 125 (CA-125), a complex pelvic mass, ascites, and carcinomatosis. These signs are not necessary for suspicion or enrollment in this protocol.
* Age > 18 years and competent to give informed consent.
* Must have a Eastern Cooperative Oncology Group (ECOG) Performance status of 0, 1, or 2 and a life-expectancy of at least 60 days.
* Adequate bone marrow function.
* Adequate renal function.
* Adequate hepatic function.
* Participants must sign an approved informed consent and authorization permitting release of personal health information.
* Women of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized.

Exclusion Criteria:

* Current use of FWGE
* Known allergy to wheat, rice (contained in the placebo), orange or the sweetener, Stevia.
* Potential participants who received neoadjuvant chemotherapy for ovarian cancer.
* An upper gastrointestinal or other condition that would impair swallowing or absorption of oral medication.
* Any serious illness or medical condition that would not permit the patient to be managed according to the protocol, including, but not to limited, any the following: History of significant neurologic or psychiatric disorder (e.g., uncontrolled psychiatric disorders) that would impair the ability to obtain consent or limit compliance with study requirement; Active uncontrolled or serious infection; Active peptic ulcer disease.
* Uncontrolled hypertension defined as systolic greater than 180 and diastolic greater than 100.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hye Sook Chon, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center March 2016 through February 2017.
Groups:
- Fermented Wheat Germ Extract (FWGE): FWGE administration 2 - 4 weeks prior to planned surgery.
- Placebo Administration: Placebo administration 2 - 4 weeks prior to planned surgery.
Period: Overall Study
Arm/Group | Fermented Wheat Germ Extract (FWGE) | Placebo Administration
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fermented Wheat Germ Extract (FWGE): FWGE administration 2-4 weeks prior to planned surgery, + Quality of Life (QoL) Surveys: FACT-O
- Placebo Administration: Placebo administration 2-4 weeks prior to planned surgery, + Quality of Life (QoL) Surveys: FACT-O
- Total: Total of all reporting groups
Arm/Group | Fermented Wheat Germ Extract (FWGE) | Placebo Administration | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 2 | 2
Age, Continuous [Median (Full Range); unit: years] | 63 [63 to 63] | 74.5 [74 to 75] | 70.6 [63 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Adverse Events Probably Related to Study Treatment
Description: Adverse events reported per treatment arm. An adverse event is the development of an untoward medical occurrence, undesirable medical condition, or recurrence or deterioration of a pre-existing medical condition subsequent to exposure to FWGE. This study will utilize the Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) for toxicity and adverse event reporting.
  Number of Adverse Events Probably Related to Study Treatment. All Adverse Events are listed, with causality noted in the Adverse Event section.
Time Frame: Up to 2 months
Population: All participants.
Measure: Number; unit: Adverse Events
Arm/Group | Fermented Wheat Germ Extract (FWGE) | Placebo Administration
Number analyzed (Participants) | 1 | 2
Adverse Events | 1 | 0

2. Secondary Outcome: Quality of Life Scores Per Treatment Arm
Description: FACT-O Quality of Life Score comparison per category and arm: Physical Well-Being; Social/Family Well-Being; Emotional Well-Being; Functional Well-Being; Additional Concerns. Score range for each question: 0 (Not at all) through 4 (Very much). High or Low Score could mean better or worse, depending on the wording of each group of questions. Investigators planned to analyze scores per treatment arm, in women who received Fermented Wheat Germ Extract (FWGE) (n=10) and those who received placebo (n=10). Drug manufacturing issues prevented investigators from completing the planned analysis.
Time Frame: Up to 2 months
Population: Drug manufacturing issues prevented investigators from completing the planned analysis.
Arm/Group | Fermented Wheat Germ Extract (FWGE) | Placebo Administration
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Level of 2,6-dimethoxy-p-benzoquinone (2,6-DMBQ)
Description: Investigators planned to perform Level comparison of 2,6-dimethoxy-p-benzoquinone (2,6-DMBQ) in the serum of women receiving FWGE versus placebo for 20 participants.
Time Frame: Up to 2 months
Population: Drug manufacturing issues prevented investigators from completing the planned analysis.
Arm/Group | Fermented Wheat Germ Extract (FWGE) | Placebo Administration
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Occurence of CA-125 Response
Description: Biomarker-based response involves assessing the participant's longitudinal CA-125 values. The definition of CA-125 response is based on the Gynecologic Cancer Intergroup (GCIG 2005) criteria. CA-125 response was to be determined and compared between FWGE and placebo treated groups of 10 participants each.
Time Frame: Up to 2 months
Population: Drug manufacturing issues prevented investigators from completing the planned analysis.
Arm/Group | Fermented Wheat Germ Extract (FWGE) | Placebo Administration
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Incidence of Changes in Tissue Proliferative Assays and Gene Expression
Description: Changes in tissue proliferative assays and gene expression per treatment arm.
Time Frame: Up to 2 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year, 1 month
Arm/Group | Fermented Wheat Germ Extract (FWGE) | Placebo Administration
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fermented Wheat Germ Extract (FWGE) (N=1) | Placebo Administration (N=2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) — Unrelated to study treatment
Investigations - Other, Total protein decreased (Investigations) | 1 (1) | 1 (1) — Unrelated to study treatment
Investigations - Other, Elevated phosphorous (Investigations) | 1 (1) | 0 (0) — Unrelated to study treatment
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Unrelated to study treatment
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Unrelated to study treatment
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) — Unrelated to study treatment
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) — Unrelated to study treatment
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) — Probably related to study treatment

LIMITATIONS AND CAVEATS:
Accrual was closed prematurely due to drug manufacturing issues and slow enrollment. Outcome Measures were designed for 20 participants, to complete a comparison of 2 study arms with 10 participants each.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT02411565/Prot_SAP_000.pdf